CLINICAL TRIAL: NCT04813874
Title: Evaluation of Maternal and Fetal Outcomes Following Nitrous Oxide and Neuraxial Labor Analgesia
Brief Title: Nitrous Oxide and Neuraxial Labor Analgesia Use on Maternal Fetal Outcomes
Acronym: NOLA
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty obtaining advanced notification of who was wanting to use nitrous
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: NOLA
Record Dates: First submitted 2017-01-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neuraxial analgesia only: Receiving neuraxial analgesia only for labor
  Interventions: Drug: Nitrous Oxide
- NO2 and neuraxial analgesia: Receiving nitrous oxide and neuraxial analgesia for labor
  Interventions: Drug: Nitrous Oxide; Procedure: Neuraxial analgesia

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous Oxide Inhalational Agent
Procedure: Neuraxial analgesia — Epidural Labor Analgesia Placement
  Other Names: Epidural placement
  Groups: NO2 and neuraxial analgesia

SUMMARY:
The purpose of this study is to evaluate maternal and neonatal outcomes in parturients who used nitrous oxide and neuraxial labor analgesia during labor.

DETAILED DESCRIPTION:
The use of nitrous oxide during labor is common in several countries including the United Kingdom, Finland, Canada, Australia and New Zealand.1, 2 The use of nitrous oxide during labor has undergone a resurgence in popularity recently in the United States and became available at Brigham and Women's hospital in August 2014.

Inhaled nitrous oxide has a rapid onset (30-50 seconds) and clearance with a half-life of about 5 minutes.3 It can be used for analgesia during the first, second and third stages of labor, as well as during post-delivery procedures such as laceration repair, manual removal of the placenta, and uterine curettage. It is also commonly used to facilitate the initiation of epidural analgesia.4 At the Brigham and Women's Hospital, a pneumatically driven gas mixer is designed to deliver a 50% oxygen and 50% nitrous oxide mixture to patients. Nitrous oxide passes readily across the placenta, and reaches equilibrium within a few minutes; the fetal maternal concentration ratio after 2 minutes of inhalation is 0.64.5 Hence, when administered at 50% concentration to the mother, the fetal concentration approximates at 32%.

Despite its long track record of maternal safety reported in numerous countries, the effect of nitrous oxide on the fetus is less well-studied. A number of studies have published data on the use of nitrous oxide for labor analgesia, including the effectiveness in labor analgesia, maternal satisfaction and maternal fetal adverse effects. Most of these studies have not identified adverse neonatal outcomes. However, these studies used Apgar scores or neonatal behavior scores as outcome measures and the quality of these studies was predominately poor.

The purpose of this study is to evaluate maternal and neonatal outcomes in parturients who used nitrous oxide and neuraxial labor analgesia during labor.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients requesting for pain relief with neuraxial analgesia and/or nitrous oxide
* health patients with no comorbidities
* singleton, vertex gestation at term

Exclusion Criteria:

* Refuse informed consent
* evidence of anticipated fetal anomalies
* significant medical or pregnancy-related diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients requesting for pain relief with neuraxial analgesia and/or nitrous oxide
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Fetal and Neonatal Outcomes | At 1 minute following birth
  Presence of Apgar Score < 7 (0-10)
Fetal and Neonatal Outcomes | At 5 minutes following birth
  Presence of Apgar Score < 7 (0-10)
Fetal and Neonatal Outcomes | At 10 minutes following birth
  Presence of Apgar Score < 7 (0-10)

SECONDARY OUTCOMES:
Maternal Outcome | During Labor at 90 minute intervals
  Visual Analogue Score (0-10)
Maternal Outcome | Any Time During Labor
  Conversion to Alternative Analgesia Method (Neuraxial or General Anesthesia)
Maternal Outcome | At Delivery
  Mode of Delivery (Vaginal or Cesarean Delivery)

IPD SHARING:
Plan to Share IPD: No